CLINICAL TRIAL: NCT07353632
Title: Re-participation for Screening-colonoscopy - Experience of colonoscpy_1
Brief Title: What Influence Re-participation in the Danish Colorectal Screening Program.
Status: Recruiting | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: OPEN, Open Patient data Explorative Network, Odense University Hospital, Region of Southern Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24/34903
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Colonoscopy; Screening Colonscopy; Pain
Keywords: Screening colonoscopy experience; Colorectal cancer screening; Patient-reported outcomes; Pain perception during colonoscopy; Screening re-participation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study investigates how participants experience screening colonoscopy within the Danish colorectal cancer screening program and how these experiences relate to clinical findings, procedural factors, and future participation in screening.

The study aims to evaluate patient-reported experiences such as pain, discomfort, preparation burden, emotional responses, and perceptions of healthcare staff, as well as staff-assessed pain during the procedure. These experiences will be examined in relation to colonoscopy findings, including polyp detection, histology, risk stratification, and colorectal cancer detection. In addition, procedure-specific variables such as insertion time, bowel preparation quality, completeness of colonoscopy, medication use, and adenoma detection rate will be analyzed in relation to patient experience.

A key focus is whether the experience of screening colonoscopy influences subsequent participation in the colorectal cancer screening program, particularly among individuals classified as low risk and re-invited for screening after two years. Registry-based follow-up will be used to assess re-participation.

Data are collected prospectively from two sources: (1) real-time procedure data entered by healthcare staff during colonoscopy and (2) patient-reported outcomes collected via a questionnaire completed shortly after the procedure. Additional outcome data are obtained from electronic medical records and national health and screening registries.

The study has no single predefined hypothesis. Instead, it serves as a data-generating platform designed to address both predefined and future research questions related to screening colonoscopy experiences, quality indicators, and screening adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing screening-derived colonoscopy as part of the Danish colorectal cancer screening program
* Written informed consent

Exclusion Criteria:

* Inability to understand or communicate in Danish
* Lack of decision-making capacity, including cognitive impairment due to dementia or brain injury
* Declines or withdraws informed consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing a screening colonoscpy
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain experienced during colonoscopy, reported by the patient | apr. 15min after colonoscopy
  11-point numerical rating scale ranging from 0 (least pain) to 10(most pain)

SECONDARY OUTCOMES:
Re-participation in screening | 2 years following colonoscopy
  2-year Re-participation rate for those calssified as low risk after index colonoscopy

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Sygehus Sønderjylland, University hospital of Southern Denmark, Aabenraa
  - Esbjerg Hospital, University Hospital of Southern Denmark, Esbjerg
  - Grindsted Sygehus, Grindsted
  - Regionshospitalet Gødstrup, Gødstrup
  - Holbæk Sygehus, Holbæk
  - Sjællands Universitetshospital Køge, Køge
  - Sjællands Universitetshospital, Nykøbing, Nykøbing Falster
  - Slagelse Sygehus, Slagelse

IPD SHARING:
Plan to Share IPD: No